CLINICAL TRIAL: NCT06328686
Title: Arginine With Whole Brain Radiation Therapy for the Treatment of Brain Metastases
Brief Title: Arginine and Whole Brain Radiation Therapy for the Treatment of Patients With Brain Metastases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Sudmeier, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005787; NCI-2023-10895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00005787 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5883-23 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-02-19; First posted 2024-03-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Arginine; Specimen Handling; Magnetic Resonance Spectroscopy; Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (IV L-arginine, WBRT) (Experimental): Patients receive L-arginine IV over 10-20 minutes followed by WBRT approximately 1 hour later for up to 10 days of treatment over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening, undergo collection of blood samples and spectroscopy on study, and undergo MRI at screening and follow up.
  Interventions: Dietary Supplement: Arginine; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Spectroscopy; Radiation: Whole-Brain Radiotherapy
- Arm B (oral L-arginine, WBRT) (Experimental): Patients receive L-arginine PO followed by WBRT approximately 1 hour later for up to 10 days of treatment over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening, undergo collection of blood samples and spectroscopy on study, and undergo MRI at screening and follow up.
  Interventions: Dietary Supplement: Arginine; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Spectroscopy; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Dietary Supplement: Arginine — Given IV or PO
  Other Names: Amino-5-guanidino-pentanoic acid; Arg; L-Arginine
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Spectroscopy — Undergo spectroscopy
Radiation: Whole-Brain Radiotherapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiation therapy

SUMMARY:
This early phase I trial evaluates different administration techniques (oral or intravenous) for arginine and tests the safety of giving arginine with whole brain radiation therapy in patients who have cancer that has spread from where it first started (primary site) to the brain (brain metastases). Arginine is an essential amino acid. Amino acids are the molecules that join together to form proteins in the body. Arginine supplementation has been shown to improve how brain metastases respond to radiation therapy. The optimal dosing of arginine for this purpose has not been determined. This study measures the level of arginine in the blood with oral and intravenous dosing at specific time intervals before and after drug administration to determine the best dosing strategy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the bioavailability of orally-administered arginine (L-arginine).

SECONDARY OBJECTIVES:

I. Test the safety of daily arginine administration with standard-fractionation whole brain radiation therapy (WBRT).

II. Determine the side effect profile of oral and intravenous (IV) L-arginine. III. Quantify frontal cortex blood volume/flow changes following L-arginine (L-arg) administration.

IV. Describe immunological effects of oral versus (vs.) IV arginine. V. Describe the metabolic effects of oral vs. IV arginine.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive L-arginine IV over 10-20 minutes followed by WBRT approximately 1 hour later for up to 10 days of treatment over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) at screening, undergo collection of blood samples and spectroscopy on study, and undergo magnetic resonance imaging (MRI) at screening and follow up.

ARM B: Patients receive L-arginine orally (PO) followed by WBRT approximately 1 hour later for up to 10 days of treatment over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening, undergo collection of blood samples and spectroscopy on study, and undergo MRI at screening and follow up.

After completion of study treatment, patients are followed up at 1 month and then quarterly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brain metastases from any primary cancer
* Planned to undergo whole-brain radiation therapy (Hippocampal avoidant is ok)
* No systemic anti-neoplastic agent concurrent with WBRT (memantine is ok)
* Not inpatient at the time of treatment start
* Age 18 or older
* Able to consent for self

Exclusion Criteria:

* Patient unwilling/unable to receive daily arginine treatment (IV or oral) for the 10 days of WBRT
* Systemic therapy continuing during WBRT
* Creatinine > 1.5 x the upper limit of normal
* Alanine aminotransferase (ALT) > 6x the upper limit of normal
* Patient planned to be treated as an inpatient
* Age < 18 years
* Adult not able to consent for self
* Pregnant
* Prisoners
* Cognitively impaired/impaired decision-making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak plasma L-arginine (arginine) and arginine metabolite concentration | Within 4 hours of oral and intravenous (IV) dosing of L-arginine
  By compartmental pharmacokinetic analysis, the plasma arginine levels at before administration, 10 min, 30 min, 1 hour, 2 hours, and 4 hours post administration will be used to estimate the median time to reach the peak plasma arginine and the mean value of peak. This will be done separately by two arms.

SECONDARY OUTCOMES:
Incidence of adverse events associated with delivering L-arginine with standard fractionation whole brain radiation therapy | At 1 week into radiation and at completion of 2 week course
  Will be evaluated using complete metabolic panel and symptom assessment. The descriptive statistics (e.g., summary statistics for numerical measurements and frequency/percentage for categorical measurements) along with data visualization (e.g., box plot repeated by time points) will mainly be considered for all 10 patients or separated by arms. As needed, the comparison between the two arms will be carried out mainly by non-parametric tests (e.g., Wilcoxon sum-rank test, Fisher's exact test). The change before and after treatment can be tested using a paired-test (e.g., Wilcoxon signed rank test). All analyses will be explored for all 10 patients or separated by arms as appropriate.
Side effect profile of oral and IV arginine | On days 1, 5, and 10
  Will be evaluated using symptom assessment at time of lab draw. The descriptive statistics (e.g., summary statistics for numerical measurements and frequency/percentage for categorical measurements) along with data visualization (e.g., box plot repeated by time points) will mainly be considered for all 10 patients or separated by arms. As needed, the comparison between the two arms will be carried out mainly by non-parametric tests (e.g., Wilcoxon sum-rank test, Fisher's exact test). The change before and after treatment can be tested using a paired-test (e.g., Wilcoxon signed rank test). All analyses will be explored for all 10 patients or separated by arms as appropriate.
Frontal cortex blood volume/flow changes with L-arginine administration | Up to 1 year
  Cerebral blood flow (CBF) and oxygen utilization will be measured using diffuse optical spectroscopy and diffuse correlation spectroscopy after arginine administration.
  The descriptive statistics (e.g., summary statistics for numerical measurements and frequency/percentage for categorical measurements) along with data visualization (e.g., box plot repeated by time points) will mainly be considered for all 10 patients or separated by arms. As needed, the comparison between the two arms will be carried out mainly by non-parametric tests (e.g., Wilcoxon sum-rank test, Fisher's exact test). The change before and after treatment can be tested using a paired-test (e.g., Wilcoxon signed rank test). All analyses will be explored for all 10 patients or separated by arms as appropriate.
Describe The Immunological Effects of Oral versus IV Arginine | Up to 10 days
  Administration of both oral and IV formulations of L-arginine will stimulate T-cell proliferation and expression of effector molecules. A phenotypic analysis of circulating immune cells will be conducted by spectral flow cytometry during treatment.
Describe The Metabolic Effects of Oral versus IV Arginine | Up to 10 days
  Administration of both oral and IV formulations of L-arginine will stimulate T-cell proliferation and expression of effector molecules. Arginine metabolites, including ornithine, citrulline, will have a delayed increase following arginine administration. A phenotypic analysis of circulating immune cells will be conducted by spectral flow cytometry during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sudmeier, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States